CLINICAL TRIAL: NCT00858104
Title: Multicentric Randomized Controlled Study of Percutaneous Laser Ablation Versus Follow Up in Benign Thyroid Nodules. Long Term Results
Brief Title: Percutaneous Laser Ablation in Benign Thyroid Nodules.Long Term Results
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Elesta S.R.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IALT-07
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Laser thermal ablation
  Interventions: Procedure: Percutaneous Laser Ablation
- 2 (No Intervention): Follow-up

INTERVENTIONS:
Procedure: Percutaneous Laser Ablation — Single session with standardized approach: Two fibers, up to 2 laser emissions; nodule volume up to 10 ml are treated by 800 Joules /ml and above 10 ml by 600 Joules/ml.The treatment is performed under local anesthesia and with diazepam sedation.
  Other Names: Arcispedale S. Maria Nuova is using commercially available system EchoLaser XVG; (Integrated Ultrasound-Laser, Elesta, Italy). Other centers are using commercially available; systems MyLab70XV (Ultrasound, Esaote, Italy) and Smart1064 BS (Nd:Yag Laser,; DEKA, Italy). Disposable Fiber Optic devices : Bare Fiber PLA THY 2111, Bare Fiber PLA S; (Asclepion Laser Technologies GmbH, Germany).
  Arms: 1

SUMMARY:
Thyroid nodule pathologies occur frequently and represent a clinical issue for the endocrinologists, surgeons, nuclear physicians as well as the general practitioners. The incidence of this pathology has been further highlighted by the introduction of the ultrasound examination into the clinical practice as 20% with impalpable thyroid nodules is now detected through ultrasound. The majority of nodules are benign and characterized by slow growth, and therefore treated with suppressive doses of levothyroxine. Long-term levothyroxine treatment has, however, several well-known side effects and limitations.

During the last years, number of controlled studies have demonstrated that ultrasound guided percutaneous laser treatment (PLA) is able to reach the target lesion within the thyroid with a high level of precision, and to destroy the thyroid tissue in a predictable and repeatable fashion, without side effects.

Aim of the study:

1. to assess 1-year and 3-year effect of laser ablation therapy on the volume of benign thyroid nodules and on nodule-related symptoms, and to compare these effects with findings in control group without active therapy;
2. to assess the eventual re-occurence of thyroid lesions (observed after other types of ablation treatment, like percutaneous ethanol injection) during a 3-year follow-up;
3. to demonstrate reproducibility of results within different environments and under different operators;
4. to validate eventual presence of major or minor side effects.

To this aim we shall randomized 200 patients either for PLA (100 pts) or standard follow-up. Patients will be recruited, treated and followed in 4 italian centers (Ospedale Regina Apostolorum - Roma, Arcispedale S. Maria Nuova - Reggio Emilia, Ospedale S. Maria della Misericordia - Perugia, Ospedale di Cisanello - Pisa) by physicians with experience in PLA.The scientific coordinator of this multicentre study is dr. Claudio Maurizio Pacella.

ELIGIBILITY:
Inclusion Criteria:

* The presence of a single nodule or dominating nodule;
* A solid or mixed echo-structure with less than 20% fluid volume;
* A lesion volume between 5 and 18 ml (greatest diameter > 3.0 cm and <= 4 cm);
* Thyroid hormone and TSH serum levels within the normalcy value;
* 2 cytologically negative examinations for suspected neoplasia (British Thyroid Association, Second class THY)within the last six months;
* Calcitonin values within the normalacy value;
* Anticoagulant treatment suspension and antiaggregation treatment suspended for at least 72 hours.

Exclusion Criteria:

* Hyperfunctioning lesion (99mTc scintigraph);
* Autoimmune thyreopathy or elevation of autoantibodies;
* Active anticoagulant treatment or antiaggregation treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Short- (1-year) and long- (3-year) term evolution of the thyroid nodules volume and symptoms after the treatment vs. simple clinical observation.(Strong Endpoint: %nodules with greater than 50% base volume reduction and %patients free of symptoms) | 3 years

SECONDARY OUTCOMES:
Assessment of short-term and long-term PLA safety, tolerability and reproducibility. | 3 years

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Azienda Ospedaliera di Perugia - Osp. S.Maria della Misericordia, Perugia, Perugia
  - Azienda Ospedaliero-Universitaria di Pisa - Presidio di Cisanello, Pisa, Pisa
  - Arcispedale S. Maria Nuova, Reggio Emilia, Reggio Emilia
  - Ospedale Regina Apostolorum, Albano Laziale, Roma

REFERENCES:
- [Background] Pacella CM, Bizzarri G, Guglielmi R, Anelli V, Bianchini A, Crescenzi A, Pacella S, Papini E. Thyroid tissue: US-guided percutaneous interstitial laser ablation-a feasibility study. Radiology. 2000 Dec;217(3):673-7. doi: 10.1148/radiology.217.3.r00dc09673. PMID 11110927
- [Background] Dossing H, Bennedbaek FN, Karstrup S, Hegedus L. Benign solitary solid cold thyroid nodules: US-guided interstitial laser photocoagulation--initial experience. Radiology. 2002 Oct;225(1):53-7. doi: 10.1148/radiol.2251011042. PMID 12354983
- [Background] Pacella CM, Bizzarri G, Spiezia S, Bianchini A, Guglielmi R, Crescenzi A, Pacella S, Toscano V, Papini E. Thyroid tissue: US-guided percutaneous laser thermal ablation. Radiology. 2004 Jul;232(1):272-80. doi: 10.1148/radiol.2321021368. Epub 2004 May 20. PMID 15155898
- [Background] Dossing H, Bennedbaek FN, Hegedus L. Effect of ultrasound-guided interstitial laser photocoagulation on benign solitary solid cold thyroid nodules - a randomised study. Eur J Endocrinol. 2005 Mar;152(3):341-5. doi: 10.1530/eje.1.01865. PMID 15757849
- [Background] Papini E, Guglielmi R, Bizzarri G, Graziano F, Bianchini A, Brufani C, Pacella S, Valle D, Pacella CM. Treatment of benign cold thyroid nodules: a randomized clinical trial of percutaneous laser ablation versus levothyroxine therapy or follow-up. Thyroid. 2007 Mar;17(3):229-35. doi: 10.1089/thy.2006.0204. PMID 17381356
- [Derived] Papini E, Rago T, Gambelunghe G, Valcavi R, Bizzarri G, Vitti P, De Feo P, Riganti F, Misischi I, Di Stasio E, Pacella CM. Long-term efficacy of ultrasound-guided laser ablation for benign solid thyroid nodules. Results of a three-year multicenter prospective randomized trial. J Clin Endocrinol Metab. 2014 Oct;99(10):3653-9. doi: 10.1210/jc.2014-1826. Epub 2014 Jul 22. PMID 25050903